CLINICAL TRIAL: NCT03792581
Title: Individualizing Mean Arterial Pressure of Head Trauma Injury Patients Using an Novel Automated System for Vasopressor Administration : a Randomized Controlled Trial
Brief Title: COntrolled MAp Trauma Brain Injury (COMAT Study)
Acronym: COMAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor was not the good one. We will redo the clincal trial gov to be concordant with the actual sponsor
Sponsor: Erasme University Hospital (Other)
Collaborators: Bicetre Hospital (Other); University of California, Irvine (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, Principal Investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A02976-49
Record Dates: First submitted 2018-12-16; First posted 2019-01-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Closed-Loop Communication
MeSH Terms: conditions — Teach-Back Communication

STUDY DESIGN:
Intervention Model Description: Manual versus automated management of MAP
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EV1000 monitor (Active Comparator): MAP management will be done as usual ( adjustment by nurses) and fluid management will be managed using the EV1000 monitoring device with the automated decision support system
  Interventions: Device: EV1000 and closed-loop system
- EV1000 monitor + closed-loop system (Experimental): fluid management will be done using the automated decision support system and MAP will be adjusted by the automated closed-loop system for vasopressor administration
  Interventions: Device: EV1000 and closed-loop system

INTERVENTIONS:
Device: EV1000 and closed-loop system — This system will recommend when patients need fluid or not and adjust vasopressor administration automatically

SUMMARY:
The goal of this randomized controlled trial will be to show that the use of a novel automated system to guide vasopressor administration in head trauma injury patients will results in more time spent with a mean arterial pressure (MAP) within the predefined MAP compared to patients managed without any automated system (manually management)

DETAILED DESCRIPTION:
In head trauma patients, the maintenance of MAP within a very narrow range is desired to avoid secondary ischemic diseases. However, the MAP needed to reach can vary over time based on intracranial pressure. Additionally, it is well know that the nurses in the Intensive care unit managed multiple patients simultaneously and cannot dedicate 100% of his-her time to adjust vasopressor infusion and/or fluid administration. Using a novel automated system can overcome this issue and may lead to more time in MAP target than the traditional management.

All patients will have the same automated system for fluid administration using the EV1000 monitoring using the AFM mode ( Assisted fluid management). This system will recommend to the clinical when to administer a fluid bolus to optimize SV and SVV. So fluid administration will be standardized in both groups. The only difference will be the management of MAP.

The goal will be to compare a treatment period of at least 3 hours during which the patient will be under continuous noradrenaline infusion. This treatment time should be within the first 48 hours of patient admission in the Intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Severe Head trauma Patients ( Glasgow score ≤8), intubated, ventilated and sedated

Exclusion Criteria:

* Glasgow score >8
* Bilateral mydriasis at the initial management

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
MEAN ARTERIAL PRESSURE (MAP) | 48 hours post-admission in the intensive care
  time when MAP will be in the predefined range (+/- 5mmHg of the predefined MAP). This target can changed over the 48 hours of patient management due to increased intracranial pressure. This target is predefined by the clinician in charge of the patient and not involved in the study.

SECONDARY OUTCOMES:
Hypotension incidence | 48 hours post-admission in the intensive care
  percentage time spent with MAP is below 5 mmHg of the predefined MAP target (hypotension) at 48 hours post admission
Hypertension incidence | 48 hours post-admission in the intensive care
  percentage time spent with MAP is above 5 mmHg of the predefined MAP target (hypotension) at 48 hours post admission
Pulsatility index | baseline (admission to the intensive care unit)
  measure of pulsatility index using the Transcranial doppler ultrasound
Pulsatility index | 24 hours post-admission to the intensive care unit
  measure of pulsatility index using the Transcranial doppler ultrasound
Pulsatility index | 48 hours post-admission to the intensive care unit
  measure of pulsatility index using the Transcranial doppler ultrasound
Mean velocity | baseline (admission to the intensive care unit)
  measure of mean velocity using the Transcranial doppler ultrasound
Mean velocity | 24 hours post-admission to the intensive care unit
  measure of mean velocity using the Transcranial doppler ultrasound
Mean velocity | 48 hours post-admission to the intensive care unit
  measure of mean velocity using the Transcranial doppler ultrasound
diastolic velocity | baseline (admission to the intensive care unit)
  measure of diastolic velocity using the Transcranial doppler ultrasound
Diastolic velocity | 24 hours post-admission to the intensive care unit
  measure of diastolic velocity using the Transcranial doppler ultrasound
Diastolic velocity | 48 hours post-admission to the intensive care unit
  measure of diastolic velocity using the Transcranial doppler ultrasound
Fluid received | 48 hours post-admission in the intensive care
  comparison of amount of fluid received during the first 48 hours post admission
Amount of vasopressor | 48 hours post-admission in the intensive care
  amount of vasopressor received during the first 48 hours post admission
Length of stay in the Intensive care unit | 30 days post-admission in the intensive care
  comparison of the length of stay in the Intensive care unit between both groups
Mean arterial pressure (MAP) | 48 hours post-admission in the intensive care
  MAP over the first 48 hours postadmission in the intensive care
Stroke volume | 48 hours post-admission in the intensive care
  stroke volume over the first 48 hours postadmission in the intensive care
cardiac index | 48 hours post-admission in the intensive care
  cardiac index over the first 48 hours postadmission in the intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Duranteau, PhD, Study Director — APHP
Locations (1):
- Joosten Alexandre, Paris, LE Kremlin Bicetre, France

IPD SHARING:
Plan to Share IPD: Undecided